CLINICAL TRIAL: NCT00894244
Title: Quantitative Evaluation of Skin Shrinkage Caused by a Non-invasive Tightening Device
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northwestern University (Other)
Responsible Party: Principal Investigator, Murad Alam, Professor in Dermatology, Otolaryngology - Head and Neck Surgery, and Surgery-Organ Transplantation, Northwestern University
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: STU1178
Record Dates: First submitted 2009-05-05; First posted 2009-05-06 (Estimated); Results first posted 2012-09-03 (Estimated); Last update posted 2021-12-28 (Actual); Status verified 2021-12

CONDITIONS: Healthy
Keywords: None- Normal healthy upper arm skin will be used.

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (1):
- Treatment (Experimental): Treatment using a non-invasive skin tightening radiofrequency device to observe skin shrinkage in the arms
  Interventions: Device: Radiofrequency device

INTERVENTIONS:
Device: Radiofrequency device — One treatment pass on one arm. 2-5 treatment passes on the other

SUMMARY:
This study is being done to measure the amount of skin shrinkage caused by a non-invasive skin tightening device.

ELIGIBILITY:
Inclusion Criteria:

* Age 30-60 y/o
* Mild to moderate laxity of arm skin
* Skin of Fitzpatrick levels I-III

Exclusion Criteria:

* Any active local arm infections
* Scarring or abnormalities in upper arm area
* Major systemic illnesses
* Any condition with delayed wound healing
* History of psychiatrist illnesses

Ages: 30 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 25 (Actual)
Dates: Start 2009-04; Primary Completion 2009-09 (Actual); Study Completion 2009-09 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Northwestern University Feinberg School of Medicine, Department of Dermatology, Chicago, Illinois, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The principal investigator will select patients presenting to the Dermatology Clinic at Northwestern Memorial Hospital who meet the inclusion criteria. These individuals will be referred to the trained researcher running the study. A brief, written description of the study will be given to the patient.
Groups:
- Thermage: Thermage ThermaCool®NXT system is a non-invasive skin tightening device designed to deliver energy to the deep dermal layer.Here it will be used to observe skin shrinkage in the arms
Period: Overall Study
Arm/Group | Thermage
Started | 25
Completed | 24
Not Completed | 1

BASELINE CHARACTERISTICS:
Arm/Group | Thermage
Number analyzed (Participants) | 25
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 20
  >=65 years | 5
Age, Continuous [Mean (Standard Deviation); unit: years] | 56 (1.78)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25
  Male | 0
Region of Enrollment [Number; unit: participants]
  United States | 25

OUTCOME MEASURES:

1. Primary Outcome: The Change in Skin Tightening in the Upper Inner or Outer Arm (as Measured by Millimeters)
Description: The documented variable was shrinkage length in millimeters as measured by the same straight ruler used throughout the experimentation. Measurements were taken immediately following treatment and thirty days following the last treatment
Time Frame: immediately following treatment and 30 days after last treatment
Measure: Number (95% Confidence Interval); unit: millimeters
Arm/Group | Thermage
Number analyzed (Participants) | 24
millimeters | 45.17 [40 to 61]

ADVERSE EVENTS:
Description: Adverse events included pain during the treatment when using the higher energy setting or treatment on the anterior, immediate erythema and swelling. However, none of the subjects experienced adverse events.
Arm/Group | Thermage
Serious Adverse Events (participants affected / at risk) | 0/25
Other Adverse Events (participants affected / at risk) | 0/25

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes